CLINICAL TRIAL: NCT01031342
Title: Early Versus Elective Colonoscopy in the Management of Lower Gastrointestinal Bleeding
Brief Title: Early Colonoscopy for Lower Gastrointestinal (GI) Bleeding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in ER rules (no longer allowed endoscopies in ER) prevented ability to perform study according to protocol
Sponsor: University of Southern California (Other)
Responsible Party: Loren Laine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-025014
Record Dates: First submitted 2009-11-02; First posted 2009-12-14 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Colonoscopy; Gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early colonoscopy (Experimental): Colonoscopy performed within 12 hours of presentation
  Interventions: Procedure: Early colonoscopy
- Elective colonoscopy (Active Comparator): Colonoscopy 36-60 hours after presentation
  Interventions: Procedure: Elective colonoscopy

INTERVENTIONS:
Procedure: Early colonoscopy — Colonoscopy within 12 hours of presentation
  Arms: Early colonoscopy
Procedure: Elective colonoscopy — Colonoscopy 36-60 hours after presentation
  Arms: Elective colonoscopy

SUMMARY:
Study hypothesis is that performing early colonoscopy in patients who present to the hospital with lower GI bleeding improves their outcome.

Patients who are admitted with bleeding from their rectum and a negative endoscopic exam of the stomach and upper intestine are randomized (like flipping a coin) to receive a colonsoscopy either as an emergency (within 12 hours) or as a routine procedure (36 hours after admission). Patients are followed during their hospitalization to see if they have further bleeding, if they require blood transfusions, if they need other diagnostic tests, if they need surgery or other treatments, and how long they stay in the hospital.

DETAILED DESCRIPTION:
The aim of this study is to determine if performing early colonoscopy in patients who present to the hospital with lower GI bleeding improves their outcome.

Patients who are admitted with bleeding from their rectum and clinical evidence of a significant bleeding episode (elevated heart rate, low blood pressure, or need for blood transfusion) have immediate upper endoscopy (examination of the stomach with a flexible rubber tube with a light and video camera on the end). If this shows no source of bleeding, the patients are randomized (like flipping a coin) to receive a colonsoscopy (examination of the large intestine with a flexible rubber tube with a light and video camera on the end) either as a emergency (within 12 hours) or as a routine procedure (36 hours after admission).

Patients are followed during their hospitalization to see if they have further bleeding, if they require blood transfusions, if they need other diagnostic tests, if they need surgery or other treatments, and how long they stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients who are admitted with rectal bleeding and one of the following high-risk features:

1. HR > 100/min
2. Systolic blood pressure <100 mmHg
3. Orthostasis -considered as increase in HR by> 20/min on assuming erect position as well as by decrease by 20 mmHg in systolic blood pressure
4. Need for blood transfusion
5. Drop in hemoglobin > 1.5 g/dl or in hematocrit of > 6% in 6 hours

Exclusion Criteria:

1. Inability to give informed consent
2. Peritoneal signs
3. Severe co-morbidities that would preclude the use of colonoscopy in standard clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Further bleeding | Duration of hospitalization (randomization to date of discharge from hospital)

SECONDARY OUTCOMES:
Diagnostic yield | Duration of hospitalization (randomization to date of discharge from hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, M.D., Principal Investigator — University of Southern California
Locations (1):
- L.A. County + U.S.C. Medical Center, Los Angeles, California, United States